CLINICAL TRIAL: NCT06253039
Title: Effects of Innovative "Living Low - Training High" Methods on Performance and Physiological Responses in Well-trained Swimmers.
Brief Title: "Living Low - Training High" Methods and Physiological Responses in Well-trained Swimmers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Collaborators: Centro de Alto Rendimento do Jamor (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RSH swimmers
Record Dates: First submitted 2023-12-21; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Normobaric Hypoxia; Hypoventilation; Normoxia
Keywords: Repeated sprint methods; Swimming performance; Training programs; V̇̇O2peak; Lactate concentration; Energetic systems; Oxygen uptake kinetics; Deoxygenation kinetics
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normobaric hypoxia (RSH) (Experimental): The RSH group will perform training sessions in a normobaric hypoxic chamber at a simulated altitude of 3000 meters (FiO2 14.5%)
  Interventions: Other: Repeated sprint
- Hypoventilation (RSH-VHL) (Experimental): RSH-VHL group will be asked to exhale down to functional residual capacity just before each repetition and then hold their breath until the end of the sprint
  Interventions: Other: Repeated sprint
- Normoxia (RSN) (Active Comparator): The control group will perform the training sessions in normoxia (FIO2, 20.9%)
  Interventions: Other: Repeated sprint

INTERVENTIONS:
Other: Repeated sprint — * The group will endure four weeks (8 sessions) of the assigned training program in addition to the regular swimming training.
  * Data collection sessions: All groups will be evaluated before and after the supervised training period in three testing sessions in normoxia separated by at least 24 hours within 7 days.
  * Training sessions: will be performed in the ski ergometer and consist of 4 sets of 5x6s all-out sprints with 24s and 5 min of passive rest between the sprints and sets, respectively.

SUMMARY:
To overcome the lack of knowledge regarding the impact of different "living low, training high" methods on swimming performance, a 4-week intervention will be carried out to determine and compare the effects of three Repeated Sprints in Hypoxia (RSH) methods with each other and with a control group. Our goal is to characterize and compare the adaptations in swimming performance and in cardiorespiratory, metabolic, and muscle oxygenation responses that can arise after a 4-week training period of RSH and RSH-voluntary hypoventilation (VHL) performed in a ski-ergometer.

DETAILED DESCRIPTION:
Recently, several new "living low training high" (LLTH) methods involving repeated sprints in hypoxia have shown promising results, especially in team sports. However, the underlying mechanisms remain mostly unclear, as does its effectiveness in improving swimming performance.

Hypoxemia can be induced by exposure to ambient hypoxia conditions, by voluntary hypoventilation at low lung volume, or by vascular occlusion (namely, blood flow restriction). Swimming performance is influenced by aerobic and anaerobic metabolism and could benefit from these different LLTH methods.

This project aims to compare the effects of repeated sprint training performed with a ski-ergometer 1) in a hypoxic chamber and 2) with voluntary hypoventilation on the performance of swimmers, as well as to characterize cardiorespiratory, metabolic, and muscle oxygenation adaptations that may contribute to the improvements achieved after four weeks of each of these types of training.

All groups will be evaluated before and after the supervised training period in three testing sessions in normoxia, separated by at least 24 hours within 7 days. Swimmers will perform: 1) time-trial (100 m front crawl) in the swimming pool to determine performance, V̇̇O2 peak, and lactate concentration following the test; 2) incremental test to exhaustion in the swim-ergometer to determine aerobic peak power, cardiorespiratory responses (V̇̇O2max, ventilatory thresholds), and maximal tissue deoxygenation; 3) time-trial test in the ski-ergometer (100 m) to access performance, muscle and pulmonary oxygen uptake kinetics, and the relative contribution of energetic systems.

Training sessions will be performed in the ski-ergometer and consist of 4 sets of 5x6s all-out sprints with 24s and 5 min of passive rest between the sprints and sets, respectively. In all testing and training sessions, pulse oxygen saturation will be measured for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Swimmers from both sexes;
* With regular participation in National Championships;
* More than five years of training experience;
* No recent exposure/acclimatization to altitude;
* No recent exposition to Blood Flow Restriction training.

Exclusion Criteria:

* athletes who had an acclimatization experience or exposure to altitude lasting more than 10 days in the last 6 months;
* pregnant or postpartum women;

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Ventilatory thresholds and maximum oxygen consumption | Before and after 4 weeks of supervised training period
  mL/kg·min
Lactate concentration | Before and after 4 weeks of supervised training period
  mmol.L-1
Muscle oximetry | Before and after 4 weeks of supervised training period
  Near-infrared spectroscopy (NIRS)
Time-trial | Before and after 4 weeks of supervised training period
  seconds

SECONDARY OUTCOMES:
Heart rate | Before and after 4 weeks of supervised training period
  bpm
Arterial oxygen saturation | Before and after 4 weeks of supervised training period
  Oxymetry (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Human Kinetics, Lisbon, Cruz-Quebrada, Portugal

IPD SHARING:
Plan to Share IPD: No